CLINICAL TRIAL: NCT05921929
Title: Safety and Pharmacokinetics of a Novel NMDA Receptor Antagonist Against Brain Related Diseases in Healthy Adult Volunteers: First-in-human, Phase I, Single Dose-escalating, Open Label Study
Brief Title: First-In-Human (FIH), Single Ascending Dose (SAD) Study of FluoroEthylNorMemantine (FENM)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: a new trial should be designed
Sponsor: ReST Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RT-IS-G-H-2301
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: PTSD; Alzheimer Disease; Brain Diseases; Neuro-Degenerative Disease; Major Depressive Disorder; Treatment Resistant Depression
Keywords: NMDA; PTSD; Alzheimer's disease; Brain Diseases; Neuro-Degenerative Disease; Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alzheimer Disease; Brain Diseases; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — fluoroethylnormemantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One single oral dose per participant (Experimental)
  Interventions: Drug: Fluoroethylnormemantine (FENM)

INTERVENTIONS:
Drug: Fluoroethylnormemantine (FENM) — Single ascending oral dose administration according to the following scheme: 20, 40, 80, 120-160, 200-240, 260-320mg/kg (six dose levels). The three upper dose levels to be administered (120-160, 200-240, 260-320mg/kg) will be precisely determined with the data collected at the end of the first three dose levels administered.

SUMMARY:
The goal of this First-In-Human (FIH) trial is to learn about safety and PharmacoKinetics (PK) in healthy adult volunteers. The main questions it aims to answer are:

* What is the safety of single ascending doses of the FluoroEthylNorMemantine (FENM)?
* What is the PK profile of single ascending doses of the FENM in human?
* What is the preliminary exploratory time course of Brain Disease Neurotrophic Factor (BDNF) plasmatic levels of single ascending doses of the FENM? Participants will receive one single oral dose of FENM.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to sign written informed consent,
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2, a total body weight >65 kg,
* efficient contraceptive mean,
* no major psychiatric disorder per the Mini-International Neuropsychiatric Interview (MINI) questionnaire,
* normal laboratory tests results, arterial Blood Pressure/pulse rate, 12-lead Electrocardiogram recording.

Exclusion Criteria:

* evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, allergic disease including drug allergies, or other severe acute or chronic medical or psychiatric condition or laboratory abnormality,
* history of febrile illness within 5 days prior to administration,
* any condition possibly affecting drug absorption,
* using of prescription drugs, vaccine, routine or as needed consumption of medications or herbal supplements,
* having positive serology, positive urine test for drugs of abuse, a general medical or psychological condition or behavior, including current substance dependence or abuse,
* history of drug or alcohol abuse within 1 year before screening,
* consuming currently of nicotine containing products, any food or any beverage containing grapefruit or grapefruit juice within 48 h prior to administration,
* having blood donation or loss of significant amount of blood within 2 months prior to study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From single dose administration to the end of the study follow-up (2 weeks later)

SECONDARY OUTCOMES:
To assess maximum plasma concentration [Cmax] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess time to Cmax [Tmax] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess minimum concentration within the dosing interval [Cmin] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess last observed plasma concentration [Clast] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess time of the minimum concentration [Tmax] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess area under the plasma concentration-time curve from 0 to the end of the dose interval [AUC 0-tau] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess area under the plasma concentration-time curve from dosing (time 0) to the time of last measured concentration [AUC 0-last] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess total area under the plasma concentration-time curve from dosing (time 0) taken to the limit as the end time becomes arbitrarily large (infinity) [AUC 0-∞] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess terminal half-life, apparent elimination half-life [T1/2] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess apparent oral clearance [CL/F] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess apparent volume of distribution [Vz/F] | At pre-dose and at 2, 4, 6, 8, 10, 12, 24, 48, 96, 189, 264 and 336hours post-dose
To assess preliminary exploratory time course of Brain Disease Neurotrophic Factor plasmatic levels of single ascending doses of the FENM | At pre-dose, at Cmax (estimated at 6-8hours post-dose) and at 48, 72 and 264hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Liège - Clinical Pharmacology Unit, Liège, Belgium